CLINICAL TRIAL: NCT00625976
Title: The Effectivity of Graded Exposure in Vivo Versus Standardized Physiotherapy in Complex Regional Pain Syndrome Type I (CRPS-I) Patients With Pain Related Fear: a Randomized Clinical Trial
Brief Title: Graded Exposure (GEXP) in Vivo Versus Physiotherapy in Complex Regional Pain Syndrome Type I (CRPS-I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 08-3-004; NL20067.068.08
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: Complex regional pain syndrome type I; Graded exposure in vivo; Physiotherapy; Pain-related fear
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Graded exposure in vivo
- 2 (Experimental)
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Graded exposure in vivo — Graded exposure in vivo according to the protocol of de Jong et al. (2005)
  Arms: 1
Behavioral: Physiotherapy — Physiotherapy according to the protocol of Oerlemans, Oostendorp, de Boo and Goris (1999)
  Arms: 2

SUMMARY:
Background:

Research on the treatment of CRPS-I, as described in the Dutch evidence based treatment guidelines (Richtlijn Complex Regional Pain Syndrome type I, 2006), mainly showed improvement at the level of pain and coping with pain. Only little improvement in functional restoration was found. Research in other pain populations such al neck- and back-pain patients has shown that pain related fear contributes to the development of functional disability. GEXP in vivo which aims on systematically reducing fear of movement, shows promising results in CRPS-I patients (de Jong et al., 2005).

Objective:

The objective of the proposed project is to compare the effectivity of GEXP in vivo with that of standardized physiotherapy in CRPS-I patients with pain related fear.

Design:

The study concerns a single blinded, single center, randomized clinical trial. The treatment will be preceded by two pre-measures. After treatment there will be one post-measurement and 3, 6 and 12 month follow-up measurements.

Population:

The study population will consist of chronic CRPS-I patients between 18 and 65, with pain related fear (PHODA-LE-score ≥ 35 and PHODA-UE-score ≥ 32).

Intervention:

The two interventions that will be compared are GEXP in vivo (de Jong et al., 2005) and standardized physiotherapy according to the protocol of Oerlemans, Oostendorp, de Boo en Goris (1999). The GEXP in vivo comprises 17 sessions of one hour, the physiotherapy treatment of 34 sessions of 30 minutes. Both treatments will be given over a period of 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis CRPS-I according to IASP criteria.
2. Pain related (PHODA-LE-score ≥ 35 and PHODA-UE-score ≥ 32)
3. Age between 18 and 65.
4. Rehabilitation treatment has been indicated.

Exclusion Criteria:

1. Pregnancy.
2. Insufficient fluency in Dutch.
3. Generalized pain syndrome.
4. Dystonia.
5. Sympathectomy of the affected extremity.
6. Psychopathology
7. Involvement in a claim regarding the disease.
8. Substance abuse.
9. Symptoms on both upper or both lower extremities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Functional disability measured with: Radboud Skills Questionnaire (RASQ; Oerlemans, Cup et al., 2000), for upper limbs; Walking Ability Questionnaire (WAQ; Perez et al., 2002), for lower limbs | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up

SECONDARY OUTCOMES:
Physical activity in daily life | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Body function and structure | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Fear of movement | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Fear of pain | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Catastrophizing Scale | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Coping with pain | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Emotional distress | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Participation | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up
Emotional involvement | 2 times pre treatment, one time post treatment and at 3, 6 and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Goossens, Dr., Principal Investigator — Maastricht University